CLINICAL TRIAL: NCT03749980
Title: MyVHL: Patient Natural History Study
Acronym: MyVHL
Status: Recruiting | Type: Observational
Sponsor: Joshua Mann, MPH (Other)
Collaborators: National Organization for Rare Disorders (Other)
Responsible Party: Sponsor-Investigator, Joshua Mann, MPH, Director of Health, VHL Alliance
Organization: VHL Alliance (Other)
Other Study IDs: 0001
Record Dates: First submitted 2018-05-30; First posted 2018-11-21 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Von Hippel-Lindau Disease; Hereditary Leiomyomatosis and Renal Cell Cancer; Birt-Hogg-Dube Syndrome; SDHB Gene Mutation
Keywords: VHL; BHD; HLRCC; SDHB; MyVHL
MeSH Terms: conditions — von Hippel-Lindau Disease; Hereditary leiomyomatosis and renal cell cancer; Birt-Hogg-Dube Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
MyVHL is a multi-patient database which helps researchers identify patterns across VHL patients. MyVHL provides you -and researchers -with more complete information about VHL, like how your lifestyle, medications, and other factors impact the disease and quality of life. These insights help you better understand the condition and help researchers know where to focus their efforts.

Due to its rarity, there is less understanding of VHL and the factors that may have an impact. The data individuals provide in MyVHL helps researchers identify and uncover factors that may increase risk, inhibit or slow tumor growth, or lead to an effective cure.

ELIGIBILITY:
Inclusion Criteria:

* All patients with von Hippel-Lindau Disease (VHL)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with von Hippel-Lindau Disease (VHL)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with CNS, kidney, adrenal, retinal, thyroid, ear, and pancreatic tumors, along with cystadenomas and lesions in the lungs, liver and skin, as they relate to VHL, BHD, HLRCC, and SDHB and specific genetic mutation. | Through study completion, an average of 1 year.
  Data regarding changes in number of CNS, kidney, adrenal, retinal, ear, and pancreatic tumors, along with cystadenomas and lesions in the lungs, liver and skin, over a lifetime.
Size of tumors in patients with CNS, kidney, adrenal, retinal, thyroid, ear, and pancreatic tumors, along with cystadenomas and lesions in the lungs, liver and skin, as they relate to VHL, BHD, HLRCC, and SDHB and specific genetic mutation. | Through study completion, an average of 1 year.
  Data regarding changes in size of CNS, kidney, adrenal, retinal, ear, and pancreatic tumors, along with cystadenomas and lesions in the lungs, liver and skin, over a lifetime.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Mann, MPH, Principal Investigator — VHL Alliance
Locations (1):
- VHL Alliance, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
When participant information is stored, the investigators are careful to protect any patient identifying information from discovery by others. Strict security safeguards are in place to reduce the chance of misuse or unplanned release of information.
  Researchers will only use participant information in a de-identified manner. De-identified means that the researchers will use participant information without knowing their identity. In some cases, they may use some identifying information about the participant for research purposes, subject to an approval process through the VHL Alliance MyVHL Research Committee. At times, the researchers will use participant information with a code, instead of their name; the code would allow results of the research to be linked back to the participant.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Larcher A, Rowe I, Belladelli F, Fallara G, Raggi D, Necchi A, Montorsi F, Capitanio U, Salonia A; OSR VHL Program. Von Hippel-Lindau disease-associated renal cell carcinoma: a call to action. Curr Opin Urol. 2022 Jan 1;32(1):31-39. doi: 10.1097/MOU.0000000000000950. PMID 34783716